CLINICAL TRIAL: NCT04410588
Title: Effect of Fentanyl With Topical Levobupivacaine With Nasal Packing in Endoscopic Nasal Surgery
Acronym: fentanyl
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa mahmoud Abd El Rady, Principal Investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: marwawael
Record Dates: First submitted 2020-05-20; First posted 2020-06-01 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-07

CONDITIONS: Analgesia During Removal of Nasal Pack After Nasal Surgery
MeSH Terms: interventions — Fentanyl; Levobupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- saline (No Intervention): saline for pain for nasal packing
- levobupivacaine (Active Comparator): levobupivacaine for pain of nasal packing
  Interventions: Drug: levobupivacaine
- fentanyl +levobupivacaine (Active Comparator): fentanyle with levobupivacaine for pain of nasal packing
  Interventions: Drug: Fentanyl + Topical Levobupivacaine

INTERVENTIONS:
Drug: Fentanyl + Topical Levobupivacaine — in nasal packing
  Arms: fentanyl +levobupivacaine
Drug: levobupivacaine — in nasal packing
  Arms: levobupivacaine

SUMMARY:
the Investigators aim to study the effect of fentanyl with topical levobupivacaine with nasal packing in endoscopic nasal surgery

ELIGIBILITY:
Inclusion Criteria:1. All patients in the age of 18-60 year 2. ASA I-II 3. Undergoing elective nasal endoscopic surgery

-

Exclusion Criteria:

1. Patients will also be excluded if any perioperative cardiovascular or respiratory event occurred which the anaesthetist with clinical responsibility for the patient thought would make the study intervention clinically unacceptable.
2. unsatisfactory preoperative peripheral arterial oxygen saturation.
3. Unsatisfactory preoperative hemoglobin level.
4. Neurological or psychiatric disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Estimated)
Dates: Start 2020-06-20 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
postoperative pain by visual analoge score | 24 houres postoperative pain assessment
  assessment of pain on removal of nasal packing after endoscopic nasal surgery by VAS score. The Visual Analogue Scale (VAS) (0, no discomfort and no pain; 10, a high level of discomfort and maximum pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Wael, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes